CLINICAL TRIAL: NCT00563953
Title: A Phase II, Open-Label, Multicenter Clinical Trial of Pegylated Liposomal Doxorubicin (Caelyx®) as Primary Treatment for Patients With Breast Cancer and a History of Heart Disease or Age Over 65 Years.
Brief Title: Caelyx as Primary Treatment for Patients With Breast Cancer and a History of Heart Disease and/or Age Over 65 Years
Acronym: CAPRICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI0702; 2007-001428-11 (EudraCT Number)
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Anthracyclines; Cardiopathy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Heart Diseases | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Primary chemotherapy regimen consisting of four cycles of pegylated-liposomal doxorubicine at 35 mg/m² IV plus CPM 600 mg/m² on Day 1 every 4 weeks followed by paclitaxel 80 mg/m²/week for 12 weeks before surgery.
  Interventions: Drug: Liposomal pegylated doxorubicine

INTERVENTIONS:
Drug: Liposomal pegylated doxorubicine — Four cycles of liposomal pegylated doxorubicine at 35 mg/m² IV combined with cyclophosphamide at 600 mg/m² on Day 1 every 4 weeks, and followed by paclitaxel 80 mg/m²/week for 12 weeks before surgery.
  Other Names: Caelyx

SUMMARY:
This is a multicenter study of a primary chemotherapy regimen in breast cancer patients at risk of developing cardiotoxicity. The aim of the study is to evaluate the response rate at surgery.

DETAILED DESCRIPTION:
This is a phase II, uncontrolled, open label, multicenter study of a primary chemotherapy regimen consisting of four cycles of liposomal pegylated doxorubicine 35 mg/m² IV plus cyclophosphamide 600 mg/m² on Day 1 every 4 weeks followed by paclitaxel 80 mg/m²/week for 12 weeks before surgery in breast cancer patients at risk of developing anthracycline-induced cardiotoxicity.

Surgery (tumorectomy, quadrantectomy, or mastectomy plus lymphadenectomy) will be performed 2 to 5 weeks after the last primary chemotherapy infusion.

Patients with > 10% of hormone receptor-positive cells will receive appropriate hormone therapy according to menopausal status.

Patients treated with breast-conserving surgery will receive radiation therapy to the mammary gland.

Patients with T4 tumors or significant axillary involvement (≥ ypN2) will receive radiation therapy to the breast or chest wall and to the lymph node chains.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer (tumor > 2 cm).
* Estrogen receptor-negative or -weakly positive tumors (less than 50% of cells), as evaluated using IHC.
* Risk factors for developing anthracycline-induced cardiomyopathy.

Exclusion Criteria:

* Severe heart failure (NYHA Class III or IV) .
* Metastatic disease.
* LVEF < 45%.
* Pregnant or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR). pCR is defined as the absence of invasive cancer in the surgical breast specimen. This definition includes evidence of carcinoma in situ only. | At surgery.

SECONDARY OUTCOMES:
Clinical response rate (complete plus partial responses). Clinical response will be assessed by imaging using the WHO criteria. | Before and after treatment with paclitaxel.
Breast-conserving surgery: tumorectomy or quadrantectomy with or without lymphadenectomy versus mastectomy. | At surgery.
Axillary node involvement after primary chemotherapy. | At surgery.
Left ventricular ejection fraction measured by echocardiography or MUGA. | At baseline, every 2 doxorubicine cycles and before surgery.
Cardiac sign/symptom questionnaire. | At baseline, every 2 doxorubicine cycles and before surgery.
Relapse-free survival at 5 years after surgery and overall survival at 5 years after study entry. | Until 5 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Gil, MD, Study Chair — Institut Català d'Oncologia
Locations (8):
- Spain (8):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Morales Meseguer, Murcia

REFERENCES:
- [Background] Gil-Gil MJ, Bellet M, Morales S, Ojeda B, Manso L, Mesia C, Garcia-Martinez E, Martinez-Janez N, Mele M, Llombart A, Pernas S, Villagrasa P, Blasco C, Baselga J. Pegylated liposomal doxorubicin plus cyclophosphamide followed by paclitaxel as primary chemotherapy in elderly or cardiotoxicity-prone patients with high-risk breast cancer: results of the phase II CAPRICE study. Breast Cancer Res Treat. 2015 Jun;151(3):597-606. doi: 10.1007/s10549-015-3415-2. Epub 2015 May 16. PMID 25981896
- [Result] Gil MJ, Bellet MC, Llombart, Ojeda B, Manso L, Mesia C, Morales S, García-Martinez H, Martínez N, Melé M, Fernández-Ortega A, Baselga J. Pegylated Liposomal Doxorubicin (PLD) as Primary Treatment in Estrogen Receptor (ER) and HER2 Poor Breast Cancer and Risk of Developing Cardiotoxicity or Elderly Patients (pt). Results from the Phase II CAPRICE Study. Cancer Research 71(24 Suppl.): 403s, 2011.(CTRC-AACR San Antonio Breast Cancer Symposium)
- [Derived] Gil-Gil MJ, Bellet M, Bergamino M, Morales S, Barnadas A, Manso L, Saura C, Fernandez-Ortega A, Garcia-Martinez E, Martinez-Janez N, Mele M, Villagrasa P, Celiz P, Perez Martin X, Ciruelos E, Pernas S. Long-Term Cardiac Safety and Survival Outcomes of Neoadjuvant Pegylated Liposomal Doxorubicin in Elderly Patients or Prone to Cardiotoxicity and Triple Negative Breast Cancer. Final Results of the Multicentre Phase II CAPRICE Study. Front Oncol. 2021 Jul 9;11:645026. doi: 10.3389/fonc.2021.645026. eCollection 2021. PMID 34307126